CLINICAL TRIAL: NCT00993980
Title: Randomized Multicenter Trial on the Effectiveness of Qigong and a Stabilizing Exercise Therapy in Patients With Low Back Pain
Brief Title: Qigong and Exercise Therapy for Low Back Pain in Adults
Acronym: QEBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QEBA-09
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Low Back Pain
Keywords: qigong; traditional chinese medicine; exercise therapy; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Qigong; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): qigong
  Interventions: Procedure: qigong
- 2 (Active Comparator): exercise therapy
  Interventions: Procedure: exercise therapy

INTERVENTIONS:
Procedure: qigong — one therapy session once a week during three months, that is 12 therapy sessions altogether
  Arms: 1
Procedure: exercise therapy — one therapy session once a week during three months, that is 12 therapy sessions altogether
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effectiveness of qigong for the treatment of low back pain compared to a stabilizing exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of chronic low back pain since at least 3 months and complaints for a maximum duration of 5 years
* low back pain more prominent than other pain in the spine
* average pain intensity of the last 7 days more or equal to 40 mm measured by a visual analogue scale (VAS 0 - 100 mm)
* intellectual and physical ability to participate in the study
* informed consent

Exclusion Criteria:

* low back pain related to malignancy
* low back pain due to an accident
* inflammatory joint disorders
* previous spine surgery
* protrusion/prolapse of a spinal disk, spondylolisthesis, with radicular symptomatology
* actually doing or planning to do other regular physical exercise during the study with possible positive effects on low back pain - such as swimming, yoga, pilates, tai chi, etc.
* planning to do another therapy during the study with possible positive effects in low back pain, such as physiotherapy, acupuncture, massage, spinal manipulation etc.
* use of pain drugs for other diseases (> 1x/week)
* pregnancy
* severe chronic or acute disease interfering with therapy attendance
* alcohol or substance abuse
* participation in another clinical trial in the last 6 months before study entry

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
average pain intensity during the last 7 days measured on a visual analogue scale (VAS) | baseline, 3, 6 and 12 months

SECONDARY OUTCOMES:
disability (Roland-Morris-Questionnaire RMQ) | baseline, 3, 6 and 12 months
health related quality of life (SF 36) | baseline, 3, 6 and 12 months
credibility of the therapy for patients | baseline, 3, 6 and 12 months
patient expectation and self efficacy | baseline, 3, 6 and 12 months
therapist's expectation | baseline, 3, 6 and 12 months
sleep quality | baseline, 3, 6 and 12 months
undesired effects | baseline, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany